CLINICAL TRIAL: NCT03476837
Title: Reducing Tobacco Exposures Among African American Socially Disadvantaged Children and Women Caregivers in the AR Delta Region
Brief Title: Reducing Tobacco Exposures Among African American Women and Children
Acronym: FRESH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Coalition for a Tobacco Free Arkansas (Unknown); Tri-County Rural Health Network (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 207306
Record Dates: First submitted 2018-02-28; First posted 2018-03-26 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Tobacco Use; Second Hand Tobacco Smoke
Keywords: secondhand smoke, African Americans, policies, tobacco use
MeSH Terms: conditions — Tobacco Use | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two groups based on the baseline assessment of CS policy (no policy/partial policy). WCGs in the treatment group will receive a three-session dose at 1, 3, and 6 months. During each treatment group session, the CHW will provide the tobacco biofeedback, motivational interviewing and educational materials at the end of the session. WCGs in the control group will receive by mail the same series of educational materials received by the treatment group at 1, 3 and 6 months. Survey and other assessments will be collected at baseline, 1, 3, 6, and 12 months.
Who Masked: Care Provider
Masking Description: The recruiter will not know the client allocation. The CHW will not know who the women are in the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Treatment (Experimental): Following baseline, the CHWs will deliver three doses of the intervention to the treatment (intervention) group over a 6-month period with follow-up at 12 months for all WCGs. At 1, 3, and 6 months, WCGs will receive motivational interviewing, educational materials and biofeedback based on the child's saliva sample and WCG's carbon monoxide.
  Interventions: Behavioral: Treatment
- Control (Active Comparator): WCGs will receive educational materials in the mail at 1, 3, and 6 months.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Treatment — The CHWs will go to the homes of the WCGs who enroll in the study and will use a culturally-adapted motivational interviewing protocol, educational messages pilot tested during the formative research phase, and biofeedback based on the child's saliva sample and WCG's carbon monoxide. Saliva samples will be collect from one child in the home at baseline and final. Baseline saliva data and carbon monoxide monitoring will be used to develop feedback that aims to motivate WCGs to implement and sustain comprehensive smoke free policies. The intervention will last 6 months. We will measure changes in primary and secondary outcomes at multiple assessment points.
  Arms: Behavioral Treatment
Behavioral: Control — Following baseline assessment, at 1, 3, and 6 months, WCGs in the control group will educational materials in the mail. Final follow-up assessments will occur at 12 months.
  Arms: Control

SUMMARY:
Secondhand smoke exposure in the home can causes sudden infant death syndrome (SIDS), asthma, respiratory illnesses, and ear infections in children. In addition to cigarette smoke, exposure to other tobacco products can further compromise the safety of children in the home. This study aims to reduce the burden of multiple tobacco exposures, improve access to preventive care, and reduce the disproportionate risk for chronic diseases, including cancer, among African American women and children living in the Arkansas Delta region. Our central hypothesis is that messages delivered by a community health worker that aim to modify knowledge, attitudes, beliefs, and subjective norms may influence the perceived threat of tobacco exposures and provide cues for African American women caregivers to implement comprehensive smokefree policies to protect their children from the harms of tobacco and in-turn, influence their quitting.

DETAILED DESCRIPTION:
Cigarette smoking among African American women in Arkansas is nearly double the prevalence for African American women in the United States. Historical trends show increasing lung cancer mortality among African American Arkansan women. Further, secondhand (SHS) exposure is highest among African Americans and persons living in poverty. Declines in SHS exposure are much slower among these groups than their comparative groups. Smokefree policies in the home can reduce SHS exposure and increase quit attempts. To date, few trials have investigated how to increase the adoption and implementation of evidence-based strategies to reduce SHS exposure in the homes of women caregivers in rural disadvantaged communities. Our study will develop and test the feasibility and efficacy of brief motivational counseling and risk-communication messages delivered by community health workers (CHWs) on the implementation of comprehensive smokefree policies (e.g. ban on cigarettes, cigars, e-cigarettes, and safekeeping of tobacco products from children) in the home. The specific aims are to 1) conduct semi-structured interviews among African American women caregivers (WCGs) and CHWs to understand risk perceptions, knowledge, attitudes, beliefs, and safety practices related to tobacco products and sociocultural and environmental influences on tobacco use and policy practices; 2) use the interview data to develop, adapt, and pilot test educational materials, motivational counseling, and tobacco exposure feedback using an iterative process of six focus groups of WCGs; and 3) assess the influence of the intervention on the primary outcome, implementation of comprehensive smokefree policies, and secondary outcomes, 7-day point prevalence abstinence and smoking reduction. H3:1 Compared to WCGs in the control group (n = 103), WCGs in the intervention group will be more likely to implement CS policies (n = 103); H3:2. will have higher 7-day point prevalence abstinence and smoke fewer cigarettes per day at 1, 3, 6, and 12 months; and H3:3. their attitudes will mediate the effects of tobacco exposure biofeedback on the outcomes. The data from this study could 1) greatly enhance the adoption of voluntary comprehensive smokefree policies in a state where the strength of state-level tobacco control policies is low and 2) reduce the risk for smoking-attributable mortality, including cancer, among socially disadvantaged women and children.

ELIGIBILITY:
Woman Caregiver Inclusion Criteria:

* African American women caregivers
* Aged 18-50
* Primary caregivers of at least one child in the home aged 6 months-14 (birth parent, guardian)
* Primary decision-maker in the AR home
* English speaking
* Can provide written informed consent
* Working phone and home address
* Smoked cigarettes and/or cigars for at least 1 year
* Low income as defined by any indicator (e.g., Medicaid; Earned Income Tax Credit; Children's Health Insurance Plan [ARKids]; subsidized housing; child care subsidies; food stamps; low-income energy assistance; free/reduced lunch program; supplemental nutrition program; Head Start program)

Woman Caregiver Exclusion Criteria:

• Women outside of intervention counties

Child Inclusion Criteria: (No longer enrolling the child bc of COVID19 and inability to collect saliva)

* Live in the home with African American WCG who is the legal parent or guardian enrolled in study
* Aged 6 months to 14 years
* Non-tobacco user

Child Exclusion Criteria:

* Child who uses any form of tobacco
* Does not live in the home of the WCG

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The caregiver must be female
Enrollment: 200 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Comprehensive smokefree policy implementation | 12 months, rolling admissions
  We will measure and compare comprehensive smoke free policy implementation in the intervention and control groups, adapting standard measures from the Tobacco Use Supplement to the Current Population Survey (i.e. "Which statement best describes rules about smoking in your home? (1) no one is allowed to smoke anywhere inside your home; (2) smoking is allowed in some places or at some time inside your home; (3) smoking is permitted anywhere inside your home")

SECONDARY OUTCOMES:
Smoking abstinence | 1, 3, 6,12 months
  We will measure 7-day point prevalence abstinence
Smoking reduction | 1, 3, 6,12 months
  We will measures number of cigarettes smoked per day

CONTACTS AND LOCATIONS:
Overall Officials: Pebbles Fagan, PhD, MPH, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones DM, Bullock S, Donald K, Cooper S, Miller W, Davis AH, Cottoms N, Orloff M, Bryant-Moore K, Guy MC, Fagan P. Factors associated with smokefree rules in the homes of Black/African American women smokers residing in low-resource rural communities. Prev Med. 2022 Dec;165(Pt B):107340. doi: 10.1016/j.ypmed.2022.107340. Epub 2022 Nov 10. PMID 36370892
- [Result] Jones DM, Kulik MC, Baezconde-Garbanati L, Bullock S, Guy MC, Fagan P. Menthol Smoking and Nicotine Dependence among Black/African American Women Smokers Living in Low-Resource, Rural Communities. Int J Environ Res Public Health. 2021 Oct 16;18(20):10877. doi: 10.3390/ijerph182010877. PMID 34682623
- [Derived] Jones DM, Clawson AH, Jin J, Bullock S, Donald K, Cooper S, Miller W, Huff Davis A, Orloff M, Bryant-Moore K, Hasan A, Guy MC, Fagan P. Evidence-based practices are effective in increasing smoke-free home rules among Black women who smoke. J Natl Cancer Inst Monogr. 2025 Aug 1;2025(70):224-234. doi: 10.1093/jncimonographs/lgaf026. PMID 40795917
- [Derived] Clawson AH, Jones DM, Bullock S, Donald K, Cottoms N, Orloff M, Fagan P. Home environment and cigarette quitting behaviors among rural Black/African American women caregivers. Health Psychol. 2025 Jan;44(1):66-79. doi: 10.1037/hea0001418. Epub 2024 Sep 30. PMID 39347763